CLINICAL TRIAL: NCT02085447
Title: A Concierge Model of Customized Adherence Enhancement Plus Long-acting Injectable Antipsychotic (CAL-C) in Individuals With Schizophrenia at Risk for Treatment Non-adherence and for Homelessness
Brief Title: A Concierge Model of CAE Plus LAI in Individuals With Schizophrenia at Risk for Treatment Non-adherence and Homelessness
Acronym: CAL-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R092670SCH4031
Record Dates: First submitted 2014-03-03; First posted 2014-03-12 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Psychotic Disorders; Schizophrenia; Schizoaffective Disorder; Medication Adherence; Medication Non-Adherence
Keywords: Homelessness; Antipsychotic Drugs; Antipsychotics; Injectables; Long Acting Injectable Antipsychotic; Psychotic Disorders; Schizophrenia; Schizoaffective Disorder; Medication Adherence; Medication Non-Adherence; Community Mental Health Centers
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Medication Adherence | interventions — Haloperidol; haloperidol decanoate; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAE-L (Experimental): Eight sessions of the manualized intervention, Customized Adherence Enhancement (CAE), will be delivered along with a long-acting injectable antipsychotic (either haloperidol decanoate or paliperidone palmitate dosed per package insert) over the course of six weeks. Study staff will also communicate with the participant's mental health provider to help ensure treatment continuation after study end.
  Interventions: Behavioral: CAE-L

INTERVENTIONS:
Behavioral: CAE-L — Eight sessions of the manualized intervention, Customized Adherence Enhancement (CAE), will be delivered along with a long-acting injectable antipsychotic (either haloperidol decanoate or paliperidone palmitate dosed per package insert) over the course of six weeks. Study staff will also communicate with the participant's mental health provider to help ensure treatment continuation after study end.
  Other Names: CAE; Customized Adherence Enhancement; LAI; Long Acting Injectable Antipsychotic; Haldol Decanoate; haloperidol decanoate; Invega Sustenna; paliperidone palmitate

SUMMARY:
This is a prospective study using a concierge model of customized adherence enhancement and long-acting injectable antipsychotic (CAL-Concierge) in 30 individuals with schizophrenia or schizoaffective disorder at risk for treatment non-adherence and for homelessness. Like the CAE-L approach, CAL-Concierge is expected to improve health outcomes among the most vulnerable of populations with schizophrenia but even more importantly, will demonstrate that it can be used to improve the efficiency and quality of care in typical practice settings.

DETAILED DESCRIPTION:
Psychotropic medications are a cornerstone of treatment for individuals with schizophrenia, but rates of full or partial non-adherence exceed 60%. There is direct correlation between non-adherence and rates of relapse in schizophrenia; on average, non-adherent patients have a risk of relapse that is 3.7 times greater than their adherent counterparts. Long-acting injectable antipsychotic (LAI) medication can improve adherence but needs to be combined with a quality behavioral program to modify long-term attitudes and behaviors.

A recently completed study funded by the Reuter Foundation and conducted by these investigators found that a novel customized psychosocial adherence enhancement intervention paired with LAI (CAE-L) reduced rates of homelessness, improved psychiatric symptoms and increased overall functioning in this very vulnerable group of individuals. CAE has been manualized and appears very acceptable to homeless people with serious mental illness. However, in spite of the very promising results, the CAE-L intervention has some important limitations that are barriers to its wide-spread future use in public health settings. These limitations are:

1. CAE-L used a PhD-level psychologist to deliver the behavioral part of the program. Many public-sector clinical settings have a very limited number of such highly trained individuals. As an alternative, social workers could be an efficient way to deliver CAE.
2. CAE-L used only haloperidol decanoate as the injectable medication. Unfortunately, akathisia-- a very distressing side effect, occurred in 40% of people. Use of a newer, better tolerated medication option could improve the investigators approach.
3. Logistic barriers preventing people who were stabilized and doing well on CAE-L to continue their improved functioning once they transitioned back to regular care settings. It is clear that there needs to be a mechanism to facilitate the successful "hand-off" of individuals who have benefitted from CAE-L into maintenance therapy. A successful transition could have substantial financial and humanitarian cost-savings.

To address these obstacles and in preparation for a large-scale randomized controlled trial of this novel, blended intervention the investigators propose to conduct a prospective study using a concierge model of customized adherence enhancement combined with a long-acting injectable antipsychotic (CAL-Concierge) in individuals with schizophrenia at risk for treatment non-adherence and for homelessness. Like the CAE-L approach, CAL-Concierge is expected to improve health outcomes among the most vulnerable of populations with schizophrenia but even more importantly, will demonstrate that it can be used to improve the efficiency and quality of care in typical practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 18 and older with schizophrenia or schizoaffective disorder as confirmed by the Mini International Psychiatric Inventory (MINI). The investigators will use a DSM-5 concordant version of the MINI if it is available at the time that the first study participant is enrolled.
* Individuals who are currently or have been recently homeless (within the past 12 months) as per revised federal definition of homelessness (Homeless Emergency Assistance and Rapid Transition to Housing. In: Development DoHaU, ed2011.)
* Known to have medication treatment adherence problems as identified by the Treatment Routines Questionnaire (TRQ, 20% or more missed medications in past week or past month)
* Ability to be rated on psychiatric rating scales.
* Willingness to take long-acting injectable medication
* Currently in treatment at a Community Mental Health Clinic (CMHC) or other treatment setting able to provide mental health care during and after study participation
* Able to provide written, informed consent to study participation.

Exclusion Criteria:

* Individuals on long-acting injectable antipsychotic medication immediately prior to study enrollment.
* Prior or current treatment with clozapine
* Medical condition or illness, which in the opinion of the research psychiatrist, would interfere with the patient's ability to participate in the trial
* Physical dependence on substances (alcohol or illicit drugs) likely to lead to withdrawal reaction during the course of the study in the clinical opinion of the treated research psychiatrist
* Immediate risk of harm to self or others
* Female who is currently pregnant or breastfeeding
* Individual who is already in permanent and supported housing that includes comprehensive mental health services (i.e. Housing First)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAE-L
Started | 30
Completed | 26
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | CAE-L
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were allowed to select as many race categories as applicable. One person selected multiple race categories: White and Hispanic.
  Participants
    Hispanic ethnicity | 2
    Caucasian | 3
    African American | 26
Region of Enrollment [Number; unit: participants]
  United States | 30
Marital Status, categorical [Count of Participants; unit: Participants]
  Single, never married | 21
  Divorced | 7
  Widowed | 1
  Missing data | 1
Type of Illness, categorical [Count of Participants; unit: Participants]
  Schizophrenia | 6
  Schizoaffective disorder | 24
Age of SMI (serious mental illness) onset, continuous [Mean (Standard Deviation); unit: years] | 19.3 (19.4)
TRQ (Tablets Routine Questionnaire) Mean, SD [Mean (Standard Deviation); unit: percentage of adherence]
  Past Week | 46.5 (35.6)
  Past Month | 43.3 (32.9)
Housing status as a percentage of the previous 180 days (%, SD) [Mean (Standard Deviation); unit: percentage of days]
  Outdoors | 6.3 (17.0)
  Short-term/emergency shelter | 13.6 (26.8)
  Transitional housing | 19.2 (30.4)
  Permanent housing with assistance | 9.0 (26.9)
  Permanent housing without assistance | 37.9 (48.2)
  Incarceration | 5.8 (15.4)
History of substance abuse (N, %) [Count of Participants; unit: Participants] | 12
History of incarceration in the last 6 months (N, %) [Count of Participants; unit: Participants] | 9
BMI (mean, SD) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index; calculated by kg/m^2
  kg/m^2 | 31.2 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tablets Routine Questionnaire (TRQ, Past Week) From Screen to Week 25 Visit
Description: The Tablets Routine Questionnaire (TRQ) determines the proportion of prescribed medication taken and is not dependent upon timing of medication provided that medication is consumed within the required day/24 hour period. This rating has demonstrated statistically significant association with past non-adherence, repeated past non-adherence, any non-adherence in the past month, and non-adherence in the past week. The TRQ format will be modified slightly to document all adherence values (an exact proportion) for each item. TRQ scores ranges from perfect adherence (0% missed) to missing all medication (100% missed). An average TRQ was calculated for individuals on more than one BD medication.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 TRQ. As such, the change from screen only calculates for those who have both values, or in this case, n=16.
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | CAE-L
Number analyzed (Participants) | 16
percentage of adherence | 56.2 (33.6)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .012, t-test, 1 sided

2. Primary Outcome: Change in Tablets Routine Questionnaire (TRQ) (Past Month) From Screen to Week 25
Description: as for outcome 1
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 TRQ. As such, the change from screen only calculates for those who have both values, or in this case, n=15.
Measure: Mean (Standard Deviation); unit: percentage of adherence
Groups:
- CAE-L: Eight sessions of the manualized intervention, Customized Adherence Enhancement (CAE), will be delivered along with a long-acting injectable antipsychotic (either haloperidol decanoate or paliperidone palmitate dosed per package insert) over the course of six weeks. Study staff will also communicate with the participant's mental health provider to help ensure treatment continuation after study end.
  CAE-L (Customized Adherence Enhancement- Long-acting injectable): Eight sessions of the manualized intervention, Customized Adherence Enhancement (CAE), will be delivered along with a long-acting injectable antipsychotic (either haloperidol decanoate or paliperidone palmitate dosed per package insert) over the course of six weeks. Study staff will also communicate with the participant's mental health provider to help ensure treatment continuation after study end.
Arm/Group | CAE-L
Number analyzed (Participants) | 15
percentage of adherence | 15.2 (26.3)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .028, t-test, 1 sided

3. Primary Outcome: Long-acting Injection (LAI) Adherence
Description: Long-acting injection (LAI) adherence will be determined as a proportion of LAI (paliperidone palmitate or haloperidol decanoate) injections received at the appropriate time (within 7 days of scheduled time).
Time Frame: Week 25
Population: There is missing data for some participants. As such, the number analyzed for LAI adherence is n=16.
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | CAE-L
Number analyzed (Participants) | 16
percentage of adherence | 90.5 (30.1)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .162, t-test, 1 sided

4. Secondary Outcome: Change in DAI (Drug Attitudes Index) From Screen to Week 25
Description: The DAI contains ten true-false items. Correct responses are scored as +1, while incorrect responses are scored as 0. The highest possible score is 10, while the lowest possible score is 0. Higher scores indicate better drug attitudes, while lower scores indicate worse drug attitudes.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 DAI. As such, the change from screen only calculates for those who have both values, or in this case, n=23.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 23
units on a scale | 8.5 (1.3)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .021, t-test, 1 sided

5. Secondary Outcome: Change in AMSQ (Attitudes Toward Mood Stabilizers Questionnaire) From Screen to Week 25
Description: The AMSQ/AMQ is used to measure attitudes towards medications. The scale contains 19 items. Responses which suggest positive attitudes towards medications are scored "0", while responses which suggest negative attitudes towards medications are scored "1". The items scores are added for a total score. Total scores range from 0 to 19. Lower total scores suggest more positive attitudes, while higher scores suggest more negative attitudes.
Time Frame: Screen, Week 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 26
units on a scale | 4.0 (2.9)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .005, t-test, 1 sided

6. Secondary Outcome: Change in PANSS (Positive and Negative Syndrome Scale; Positive Symptoms Scale) From Screen to Week 25
Description: The PANSS is used to assess patients for positive and negative symptoms of schizophrenia or schizoaffective disorder. The Positive Symptoms Subscale consists of 7 questions. Each item is rated on a scale of 1 (Absent) to 7 (Extreme). Total scores for the Positive Symptoms Subscale range from 7-49. Higher scores indicate more symptoms of psychopathology. There is no aggregate score for this measure, as the subscales are to be scored separately.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 PANSS. As such, the change from screen only calculates for those who have both values, or in this case, n=24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 24
units on a scale | 21.2 (5.3)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p < .001, t-test, 1 sided

7. Secondary Outcome: Change in PANSS (Positive and Negative Syndrome Scale; Negative Symptoms Scale) From Screen to Week 25
Description: The PANSS is used to assess patients for positive and negative symptoms of schizophrenia or schizoaffective disorder. The Negative Symptoms Subscale consists of 7 questions. Each item is rated on a scale of 1 (Absent) to 7 (Extreme). Total scores for the Negative Symptoms Subscale range from 7-49. Higher scores indicate more symptoms of psychopathology. There is no aggregate score for this measure, as the subscales are to be scored separately.
Time Frame: Screen, Week 25
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 24
units on a scale | 12.1 (6.1)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .197, t-test, 1 sided

8. Secondary Outcome: Change in PANSS (Positive and Negative Syndrome Scale; Composite Scale) From Screen to Week 25
Description: The PANSS is used to assess patients for positive and negative symptoms of schizophrenia or schizoaffective disorder. The Composite Scale is scored by subtracting the negative score from the positive score. This yields a bipolar index that ranges from -42 to +42. The bipolar composite scale simply expresses the direction and magnitude of difference between positive and negative syndromes. Scores >0 indicate there are more positive symptoms of schizophrenia endorsed, and scores <0 indicate there are more negative symptoms of schizophrenia endorsed. There is no aggregate score for this measure, as the subscales are to be scored separately.
Time Frame: Screen, Week 25
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 24
units on a scale | .8 (6.6)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p < .001, t-test, 1 sided

9. Secondary Outcome: Change in PANSS (Positive and Negative Syndrome Scale; General Psychopathology) From Screen to Week 25
Description: The PANSS is used to assess patients for positive and negative symptoms of schizophrenia or schizoaffective disorder. The General Psychopathology Subscale consists of 16 questions. Each item is rated on a scale of 1 (Absent) to 7 (Extreme). Total scores range from 16-112 on the General Psychopathology scale. Higher scores indicate more symptoms of psychopathology. There is no aggregate score for this measure, as the subscales are to be scored separately.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 PANSS. As such, the change from screen only calculates for those who have both values, or in this case, n=22.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 22
units on a scale | 24.7 (6.4)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p < .001, t-test, 1 sided

10. Secondary Outcome: Change in CGI (Clinical Global Impression) From Screen to Week 25
Description: The CGI evaluates global psychopathology illness severity on a 7 point Likert Scale (minimum score = 1; maximum score = 7) with higher scores indicating worse pathology.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 CGI. As such, the change from screen only calculates for those who have both values, or in this case, n=22.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 22
units on a scale | 2.9 (.8)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p < .001, t-test, 1 sided

11. Secondary Outcome: Change in ASSIST GRS (Alcohol, Smoking and Substance Involvement Screening Test ) From Screen to Week 25
Description: The ASSIST was used to measure drug use. A total score is derived by combining item scores (minimum score = 0; maximum score = 382). Higher scores indicate higher risk of lifestyle problems, including health.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 ASSIST. As such, the change from screen only calculates for those who have both values, or in this case, n=20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | 2.0 (2.5)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .053, t-test, 1 sided

12. Secondary Outcome: Change in SOFAS (Social and Occupational Functioning Assessment Scale) From Screen to Week 25
Description: Evaluates social and occupational functioning on a scale of 0 (Inadequate information) to 100 (Superior functioning). It is a one-item measure.
Time Frame: Screen, Week 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 26
units on a scale | 63.1 (8.7)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p < .001, t-test, 1 sided

13. Secondary Outcome: Change in AIMS (Abnormal Involuntary Movement Scale) From Baseline to Week 25
Description: The AIMS is used to monitor for the development of involuntary movements that may occur as a result of certain psychotropic medication. It contains 14 items, 10 of which are rated on a scale of 0 (None) to 4 (Severe). The remaining four items are "yes or no" questions. Items 1 thru 7 are added for a total score, while item 8 is used as an overall severity index. Total scores range from 0 to 28. Higher scores indicate more adverse outcomes.Items 9 thru 12 provide additional information that may be useful in determining lip, jaw, and tongue movements.
Time Frame: Baseline, Week 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 23
units on a scale | 1.5 (2.5)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .821, t-test, 1 sided

14. Secondary Outcome: Change in SAS (Simpson Angus Scale) From Screen to Week 25
Description: The Simpson-Angus Scale is used to monitor for neurological and musculoskeletal side effects that may be a result of certain psychotropic medications. The scale consists of 10 questions which each can be rated on a scale of 0 to 4. Scores for each item are added to produce a total score. Total scores range from 0 to 40. Higher scores indicate more adverse outcomes.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 SAS. As such, the change from screen only calculates for those who have both values, or in this case, n=20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | 0.0 (0.2)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .330, t-test, 1 sided

15. Secondary Outcome: Change in BARS (Barnes Akathisia Rating Scale) From Screen to Week 25
Description: This scale is used to measure the presence of akathisia, as may result from use of certain psychotropic medications. The scale contains four items and the score for each item is added to produce the total score. Total scores range from 0 to 14. Higher scores indicate more adverse outcomes.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 BARS. As such, the change from screen only calculates for those who have both values, or in this case, n=20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | .3 (1.3)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .425, t-test, 1 sided

16. Secondary Outcome: Change in ESRS-A (Extrapyramidal Symptoms Scale-Abbreviated; Parkinsonism) From Screen to Week 25
Description: For the subjective examination scoring is on a 4-point scale (0=Absent;1=Mild, 2=Moderate, 3=Severe). The evaluator takes into account the verbal report of the patient on: 1) the frequency and duration of the symptom during the day; 2) the number of days the symptom was present during the last week; and, 3) the subjective evaluation of the intensity of the symptom by the patient. The score for Parkinsonism (including akathisia), ranges from 0 to 102 (17 items), and is based on all items of the Parkinsonism examination: tremor (0-48), gait and posture (0-6), postural stability (0-6), rigidity (0-24), expressive automatic movements (0-6), bradykinesia (0-6), akathisia (0-6). Higher scores indicate more severity.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 ESRS-A. As such, the change from screen only calculates for those who have both values, or in this case, n=20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | 0.0 (0.2)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .577, t-test, 1 sided

17. Secondary Outcome: Change in ESRS-A (Extrapyramidal Symptoms Scale-Abbreviated; Dystonia) From Screen to Week 25
Description: For the subjective examination scoring is on a 4-point scale (0=Absent;1=Mild, 2=Moderate, 3=Severe). The evaluator takes into account the verbal report of the patient on: 1) the frequency and duration of the symptom during the day; 2) the number of days the symptom was present during the last week; and, 3) the subjective evaluation of the intensity of the symptom by the patient. The score for dystonia ranges from 0 to 60 (10 items), and is formed by including both acute and chronic dystonia, based on the dystonia examination. Higher scores indicate more severity.
Time Frame: Screen, Week 25
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | 0.0 (0.0)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .330, t-test, 1 sided

18. Secondary Outcome: Change in ESRS-A (Extrapyramidal Symptoms Scale-Abbreviated; Dyskinesia) From Screen to Week 25
Description: For the subjective examination scoring is on a 4-point scale (0=Absent;1=Mild, 2=Moderate, 3=Severe). The evaluator takes into account the verbal report of the patient on: 1) the frequency and duration of the symptom during the day; 2) the number of days the symptom was present during the last week; and, 3) the subjective evaluation of the intensity of the symptom by the patient. Score for TD, ranging from 0 to 42, is based on the sum of all seven items in the TD objective examination. Higher scores indicate more severe symptomology.
Time Frame: Screen, Week 25
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | 1.4 (2.2)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .706, t-test, 1 sided

19. Secondary Outcome: Change in ESRS-A (Extrapyramidal Symptoms Scale-Abbreviated; Akathisia)
Description: For the subjective examination scoring is on a 4-point scale (0=Absent;1=Mild, 2=Moderate, 3=Severe). The evaluator takes into account the verbal report of the patient on: 1) the frequency and duration of the symptom during the day; 2) the number of days the symptom was present during the last week; and, 3) the subjective evaluation of the intensity of the symptom by the patient. The score for akathisia is separated from the Parkinsonism score and is based on the combined score of subjective akathisia (item 6 of the questionnaire) and objective akathisia (item 7 of the Parkinsonism/Akathisia objective examination). This subscore total ranges from 0 to 6. Higher scores indicate more severity.
Time Frame: Screen, Week 25
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 20
units on a scale | .2 (.9)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .481, t-test, 1 sided

20. Secondary Outcome: Change in Hospitalizations (Psychiatric) in the Past 6 Months From Screen and Week 25
Description: Change in number of psychiatric hospitalizations from the past 6 months from Screen and Week 25. This is calculated by subtracting the number of psychiatric hospitalizations at screen from the number of psychiatric hospitalizations at week 25.
Time Frame: Screen, Week 25
Measure: Mean (Standard Deviation); unit: hospital visits
Arm/Group | CAE-L
Number analyzed (Participants) | 26
hospital visits | .2 (.4)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .020, t-test, 1 sided

21. Secondary Outcome: Change in Hospitalizations (Medical) in the Past 6 Months From Screen and Week 25
Description: as for outcome 20
Time Frame: Screen, Week 25
Measure: Mean (Standard Deviation); unit: hospital visits
Arm/Group | CAE-L
Number analyzed (Participants) | 26
hospital visits | .2 (.4)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .103, t-test, 1 sided

22. Secondary Outcome: Percentage Change of Days of Sub-optimal Housing in the Past Six Months; Change From Screen to Week 25
Description: Change in number of sub-optimal housing from the past 6 months from Screen and Week 25. This is calculated by subtracting the percent of sub-optimal housing at screen from the number of sub-optimal housing at week 25.
Time Frame: Screen, Week 25
Population: There is missing data for some participants on the week 25 housing status. As such, the change from screen only calculates for those who have both values, or in this case, n=20.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | CAE-L
Number analyzed (Participants) | 20
percentage of days | 29.0 (38.2)
Statistical Analysis 1: Comparison: CAE-L; Test type: Superiority; p = .063, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CAE-L
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAE-L (N=30)
psychiatric hospitalization due to suicidal ideation (Psychiatric disorders) | 1 (1)
hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
frostbite (Infections and infestations) | 1 (1)
spider bite (Infections and infestations) | 1 (1)
acute alcoholic hepatitis (Hepatobiliary disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No